CLINICAL TRIAL: NCT03326830
Title: Prehospital High-Flow Nasal Oxygen Therapy in Patients With Acute Hypoxemic Respiratory Failure: A Randomized, Open-label, Bi-center, Pilot Study
Brief Title: Prehospital High-Flow Nasal Oxygen Therapy
Acronym: PRHOXY-1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Régional d'Orléans (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHRO-2017-09; 2017-A01922-51 (Other: IDRCB number issued by the French Government); CHRO-2017-09 (Other: Study code issued by the sponsor)
Record Dates: First submitted 2017-10-27; First posted 2017-10-31 (Actual); Last update posted 2023-02-17 (Actual); Status verified 2023-02

CONDITIONS: Acute Respiratory Failure With Hypoxia; Oxygen Inhalation Therapy; Prehospital Setting
Keywords: Respiratory Insufficiency; Oxygen Inhalation Therapy
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Intervention Model Description: Bi-center, open-label, parallel, randomized trial with 1:2 allocation ratio (2 patients assigned to standard oxygen therapy for 1 patient assigned to High Flow Nasal Oxygen therapy)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard oxygen therapy (Active Comparator): Standard oxygen therapy will be delivered using any device or combination of devices that are part of usual care: nasal oxygen, and mask with or without a reservoir bag and with or without the Venturi system. The flow will be tapered to target an SpO2 ≥ 95%
  Interventions: Device: Standard oxygen therapy
- High-flow nasal oxygen (HFNO) (Experimental): Experimental: High-flow nasal oxygen (HFNO) group Device that delivers humidified and warmed high-flow oxygen at flows between 30-60L/min HFNO will be initiated at a flow rate between 30-60 L/min and FiO2 titrated for a target of SpO2 ≥ 95%.
  Interventions: Device: High-flow nasal oxygen

INTERVENTIONS:
Device: High-flow nasal oxygen — oxygen therapy will be delivered through a dedicated system, the Airvo2™ (Fisher&Paykel, New-Zealand).
  Arms: High-flow nasal oxygen (HFNO)
Device: Standard oxygen therapy — Oxygen therapy will be delivered using standard devices such as nasal canula or face mask with or without rebreathing bag
  Arms: Standard oxygen therapy

SUMMARY:
The purpose of the present project is to compare High-Flow Nasal Oxygen therapy with Standard Oxygen therapy, initiated in the prehospital setting in patients with acute hypoxemia respiratory failure, in terms of oxygenation at arrival to the hospital and need of mechanical ventilation during the subsequent 28 days

DETAILED DESCRIPTION:
Patients with respiratory distress and an SpO2 below 90% in the prehospital setting will be randomized to receive either high-flow nasal oxygen therapy through a dedicated device or standard oxygen therapy through standard devices such as nasal cannula or face mask. Need of mechanical ventilation either invasive or noninvasive from enrollment to day 28 and time course of oxygenation between first SpO2 measured on scene and arrival to the hospital will be the main outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* First SpO2 on scene <90%
* At least one other sign of respiratory distress defined by (a) respiratory distress with a respiratory rate ≥ 25/min; (b) laboured breathing
* No advance directives or known decisions of Do Not intubate or Do Not Ventilate order.

Exclusion Criteria:

* Known COPD or other hypercapnic chronic respiratory failure
* age <18 years
* Pregnancy or breastfeeding
* Anatomical factors precluding the use of a nasal cannula
* Emergency intubation required
* Patients with tracheostomy
* Patient transported to a hospital not involved in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2017-12-21 (Actual); Primary Completion 2022-08-10 (Actual); Study Completion 2022-08-10 (Actual)

PRIMARY OUTCOMES:
need of mechanical ventilation | 28 days
  cumulative incidence of the use of tracheal intubation or noninvasive ventilation (whichever comes first) from enrolment to day 28

SECONDARY OUTCOMES:
Hypoxemia | 1 hour
  Frequency of hypoxemia, defined as sustained (at least 5 min) SpO2 below 90% (SpO2 will be continuously recorded throughout the prehospital medical care period) from the beginning of the intervention period until arrival at Emergency Department or other hospital ward.
Severe hypoxemia | 1 hour
  Frequency of severe hypoxemia, defined as sustained (at least 5 min) SpO2 below 85% from the beginning of the intervention period until arrival at Emergency Department or other hospital ward.
Survival | 28 days
  Probability of survival from inclusion to day 28
SpO2 | 1 hour
  Time course of SpO2
Respiratory rate | 1 hour
  Time course of respiratory rate
Heart rate | 1 hour
  Time course of heart rate
Tracheal intubation | 28 days
  Cumulative incidence of tracheal intubation from inclusion to day 28.
Noninvasive ventilation | 28 days
  Cumulative incidence of noninvasive ventilation use for acute respiratory failure from inclusion to day 28
arterial pH | 1 hour
  arterial pH (units) measured at hospital arrival
arterial PaCO2 | 1 hour
  arterial PaCO2 (mmHg) measured at hospital arrival
arterial PaO2 | 1 hour
  arterial PaO2 (mmHg) measured at hospital arrival
Dyspnea | 1 hour
  Dyspnea intensity as assessed by the patient him/herself at hospital arrival using the following dyspnea score: frank improvement: +2; mild improvement: +1; No change: 0; slight worsening: -1; frank worsening:-2.
Serious Adverse Events | Day 28
  The number of serious adverse events during the intervention phase of the study

CONTACTS AND LOCATIONS:
Overall Officials: Mai-Anh Nay, MD, Principal Investigator — Centre Hospitalier Régional d'Orléans
Locations (2):
- France (2):
  - CHR d'ORLEANS, Orléans
  - Brigade des Sapeurs Pompiers de Paris, Paris

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Prekker ME, Feemster LC, Hough CL, Carlbom D, Crothers K, Au DH, Rea TD, Seymour CW. The epidemiology and outcome of prehospital respiratory distress. Acad Emerg Med. 2014 May;21(5):543-50. doi: 10.1111/acem.12380. PMID 24842506
- [Background] Kelly AM, Holdgate A, Keijzers G, Klim S, Graham CA, Craig S, Kuan WS, Jones P, Lawoko C, Laribi S; AANZDEM study group. Epidemiology, prehospital care and outcomes of patients arriving by ambulance with dyspnoea: an observational study. Scand J Trauma Resusc Emerg Med. 2016 Sep 22;24(1):113. doi: 10.1186/s13049-016-0305-5. PMID 27658711
- [Background] Stiell IG, Spaite DW, Field B, Nesbitt LP, Munkley D, Maloney J, Dreyer J, Toohey LL, Campeau T, Dagnone E, Lyver M, Wells GA; OPALS Study Group. Advanced life support for out-of-hospital respiratory distress. N Engl J Med. 2007 May 24;356(21):2156-64. doi: 10.1056/NEJMoa060334. PMID 17522399
- [Background] Fontanari P, Burnet H, Zattara-Hartmann MC, Jammes Y. Changes in airway resistance induced by nasal inhalation of cold dry, dry, or moist air in normal individuals. J Appl Physiol (1985). 1996 Oct;81(4):1739-43. doi: 10.1152/jappl.1996.81.4.1739. PMID 8904594
- [Background] Sim MA, Dean P, Kinsella J, Black R, Carter R, Hughes M. Performance of oxygen delivery devices when the breathing pattern of respiratory failure is simulated. Anaesthesia. 2008 Sep;63(9):938-40. doi: 10.1111/j.1365-2044.2008.05536.x. Epub 2008 Jun 6. PMID 18540928
- [Background] Li J, Fink JB, Ehrmann S. High-flow nasal cannula for COVID-19 patients: low risk of bio-aerosol dispersion. Eur Respir J. 2020 May 14;55(5):2000892. doi: 10.1183/13993003.00892-2020. Print 2020 May. PMID 32299867
- [Background] Leonard S, Strasser W, Whittle JS, Volakis LI, DeBellis RJ, Prichard R, Atwood CW Jr, Dungan GC 2nd. Reducing aerosol dispersion by high flow therapy in COVID-19: High resolution computational fluid dynamics simulations of particle behavior during high velocity nasal insufflation with a simple surgical mask. J Am Coll Emerg Physicians Open. 2020 Jun 11;1(4):578-591. doi: 10.1002/emp2.12158. eCollection 2020 Aug. PMID 32838373